CLINICAL TRIAL: NCT03496974
Title: A Phase II, Open Label, Dose Escalation Study of Bermekimab (MABp1) in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Phase II Study of Bermekimab (MABp1) in Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-PT044
Record Dates: First submitted 2018-04-04; First posted 2018-04-12 (Actual); Results first posted 2019-07-30 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: 200 mg cohort (Experimental): The dose of bermekimab for Group A is 200 mg (2ml of the 100 mg/ml formulation)
  Interventions: Drug: Bermekimab Monoclonal Antibody 200 mg
- Group B: 400 mg cohort (Experimental): The dose of bermekimab for Group B is 400 mg (2ml of the 200 mg/ml formulation) administered weekly by subcutaneous injection
  Interventions: Drug: Bermekimab Monoclonal Antibody 400 mg

INTERVENTIONS:
Drug: Bermekimab Monoclonal Antibody 200 mg — 200 mg subcutaneous injection
  Arms: Group A: 200 mg cohort
Drug: Bermekimab Monoclonal Antibody 400 mg — 400 mg subcutaneous injection
  Arms: Group B: 400 mg cohort

SUMMARY:
A Phase 2 study of Bermekimab (MABp1) in patients with atopic dermatitis.

DETAILED DESCRIPTION:
A Phase 2, Open Label, Dose Escalation Study of Bermekimab (MABp1) in Patients with Moderate to Severe Atopic Dermatitis. The study is multi center and will consist of two dose levels:

Group A (n=9): patients will receive a total of 4 x 200mg subcutaneous injections of bermekimab. Dosing will occur weekly from visit 1 to visit 4, inclusive.

Group B (n=20): patients will receive a total of 8 x 400 mg subcutaneous injections of bermedimkb. Dosing will occur weekly from visit 1 to visit 8, inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided by the patient
* Age 18 years or greater
* Chronic Atopic Dermatitis present for at least 3 years
* Disease is not responsive to topical medications, or for whom topical treatments are not indicated or desired.
* Willing and able to comply with all clinic visits and study-related procedures
* EASI score ≥16 at screening and baseline visits
* IGA score ≥3 at screening and baseline visits
* ≥10% body surface area (BSA) of AD involvement at screening and baseline visits
* Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable or undesired.

Exclusion Criteria:

* Treatment with an investigational drug within 8 weeks of baseline visit
* Having received the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment:

  1. Immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  2. Phototherapy for AD
* Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week before the baseline visit
* Initiation of treatment during the screening period with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (patients may continue using stable doses of such moisturizers if initiated before the screening visit)
* Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit.
* History of severe allergic or anaphylactic reactions to monoclonal antibodies.
* Administration of any live (attenuated) vaccine within 4 weeks prior to the baseline.
* Any history of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell carcinoma, basal cell carcinoma or localized carcinoma in situ of the cervix
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. NOTE: patients may be rescreened after infection resolves
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (eg, tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening
* Positive with hepatitis B surface antigen (HBsAg) or hepatitis C antibody at the screening visit
* Presence of skin comorbidities that may interfere with study assessments
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study. Examples include, but are not limited to, patients with short life expectancy, patients with uncontrolled diabetes (HbA1c ≥ 9%), patients with cardiovascular conditions (eg, stage III or IV cardiac failure according to the New York Heart Association classification), severe renal conditions (eg, patients on dialysis), hepato-biliary conditions (eg, Child-Pugh class B or C), neurological conditions (eg, demyelinating diseases), active major autoimmune diseases (eg, lupus, inflammatory bowel disease, rheumatoid arthritis, etc.), other severe endocrinological, gastrointestinal, metabolic, pulmonary or lymphatic diseases. The specific justification for patients excluded under this criterion will be noted in study documents (chart notes, case report forms [CRFs], etc.)
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study
* Where relevant, women unwilling to use adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Centers Research & Education, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 mg Cohort: Bermekimab Monoclonal Antibody 200 mg: 200 mg subcutaneous injection
- 400 mg Cohort: Bermekimab Monoclonal Antibody 400 mg: 400 mg subcutaneous injection
Period: Overall Study
Arm/Group | 200 mg Cohort | 400 mg Cohort
Started | 10 | 28
Completed | 9 | 20
Not Completed | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort | Total
Number analyzed (Participants) | 10 | 28 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 22 | 30
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (16.78) | 48.54 (19.14) | 47.92 (18.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 25
  Male | 3 | 10 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 5 | 26 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 78.2 (23.34) | 74.76 (16.4) | 75.66 (18.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs)
Description: Safety and tolerability endpoints were evaluated by monitoring all the adverse events from clinical and laboratory reporting, vital signs, physical examinations, ECG and urinalysis. All the Adverse Events that the subjects experienced from Visit 1 Day 1 (Post-injection) until 7 days after the last administration of the study drug were captured in the clinical database. AEs are coded using medical dictionary - MedDRA Version 21.0 and the severity was assigned using CTCAE version 4.03.
Time Frame: From Visit 1 (Post-injection) until 7 days after the last administration of the study drug.
Population: All subjects who have received at least one dose of bermekimab were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
Participants | 3 | 6

2. Secondary Outcome: Change in Eczema Area and Severity Index (EASI) Score, From Baseline to Week 7 (or Last Visit)
Description: EASI score will assess severity and extent of AD with respect to erythema, excoriation, infiltration and lichenification at 4 anatomic sites of the body: lower and upper extremities, trunk and head. The total EASI score shall be in a range of 0 to 72 points (from no disease to maximum disease severity, respectively).
  Group A: Change= (Baseline - Week 4 score); Group B: Change= (Baseline - Week 7 score)
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with EASI score assessment at specified time-points. Missing values imputed by last observation carried forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 28.18 [20.16 to 36.2] | 29.79 [26.38 to 33.2]
  Week 4/ Week 7 | 22.73 [12.61 to 32.85] | 7.35 [4.56 to 10.14]
  Change | 5.45 [-1.85 to 12.75] | 22.44 [17.75 to 27.13]

3. Secondary Outcome: Pharmacokinetics (PK) Assessment at Week 7
Description: An enzyme-linked immunosorbent assay (ELISA) has been developed to specifically measure bermekimab levels in human plasma. Blood will be drawn into a single 6 ml Na-Heparin collection tube at each PK collection time point. These samples will be collected per the study lab manual and immediately shipped to the Sponsor for PK analysis. The PK samples will also be used to test for the presence of antibodies against bermekimab.
  PK sample collection time points are as follows:
  Group A: Pre-dose at visits 1-5; visit 5 is reported Group B: Pre-dose at visit 1, visit 3, visit 5 and visit 8; visit 8 is reported
Time Frame: Group A: Week 4; Group B: Week 7
Population: Number of participants analyzed = participants with pk analysis data at specified time-point. Missing values were not included in this analysis.
Measure: Mean (95% Confidence Interval); unit: (μg/mL)
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 6 | 22
(μg/mL) | 12.6 [9.7 to 15.5] | 47.1 [36.7 to 57.6]

4. Secondary Outcome: Number of Patients Achieving Investigator's Global Assessment (IGA) Response (0 or 1) at Week 7
Description: IGA assesses disease severity and clinical response using a 5-point scale: 0 = clear, 1= almost clear, 2 = mild, 3 = moderate, 4 = severe. The score is determined by ranking the extent of erythema and population/infiltration. A clinical response to therapy will be an IGA score of 0 (clear) or 1 (almost clear). Patients receiving more than one treatment with additional medication for AD exacerbation during the study or who are missing IGA scores at visit 8 (week 7) will be treated as non-responders. For the 200 mg group, IGA was recorded at visits 1,3, and 5; visit 5 is reported. For the 400 mg group, IGA was recorded at visits 1-8, visit 8 was reported.
Time Frame: Group A: Week 4; Group B: Week 7
Population: All subjects who have received at least one dose of bermekimab were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
Participants | 0 | 7

5. Secondary Outcome: Number of Patients Achieving ≥2 IGA Score Reduction at Week 7
Description: IGA assesses disease severity and clinical response using a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe. The score is determined by ranking the extent of erythema and papulation/infiltration. A clinical response to therapy will be an IGA score of 0 (clear) or 1 (almost clear).
Time Frame: Group A: Week 4; Group B: Week 7
Population: Number of participants analyzed = participants with IGA score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
Participants | 1 | 11

6. Secondary Outcome: Change in Peak Weekly Averaged Pruritus Numerical Rating Scores (Overall Itch) From Baseline to Week 7
Description: The NRS rating system captures the intensity of patient's itch, both maximum and average intensity over a 24-hour period. The following question was presented to patients: "How would you rate your itch at the worst moment and on average during the previous 24 hours a scale of 0-10 (0=no itch and 10=worst possible itch)?
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with pruritus NRS score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 6.50 [4.56 to 8.44] | 7.91 [7.51 to 8.3]
  Week 4/ Week 7 | 3.66 [1.48 to 5.84] | 2.51 [1.44 to 3.59]
  Change | 2.84 [0.65 to 5.03] | 5.4 [4.32 to 6.47]

7. Secondary Outcome: Change in Peak Weekly Averaged Pruritus Numerical Rating Scores (Worst Moment Itch) From Baseline to Week 7
Description: as for outcome 6
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 6.8 [4.59 to 9.01] | 7.96 [7.42 to 8.51]
  Week 4/ Week 7 | 3.71 [1.54 to 5.88] | 2.34 [1.33 to 3.36]
  Change | 3.09 [0.64 to 5.54] | 5.62 [4.55 to 6.69]

8. Secondary Outcome: Change in SCORing Atopic Dermatitis (SCORAD) Score From Baseline to Week 7
Description: SCORAD was developed by the European Task Force on Atopic Dermatitis. (Severity scoring of Atopic Dermatitis: the SCORAD index), as a measure of disease severity in AD. It includes assessment of the eczema in addition to patient-reported symptoms. Total score ranges from 0 to 103 (no disease to most severe disease, respectively).
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with SCORAD score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 59.44 [51.6 to 67.27] | 70.80 [65.93 to 75.67]
  Week 4/ Week 7 | 48.4 [36.49 to 60.3] | 26.10 [18.56 to 33.63]
  Change | 11.04 [0.36 to 21.71] | 44.70 [35.88 to 53.53]

9. Secondary Outcome: Number of Patients Achieving 50% or Greater Reduction in EASI Score at Week 7
Description: EASI score will assess severity and extent of AD with respect to erythema, excoriation, infiltration and lichenification at 4 anatomic sites of the body: lower and upper extremities, trunk and head. The total EASI score shall be in a range of 0 to 72 points (from no disease to maximum disease severity, respectively).
Time Frame: Group A: Week 4; Group B: Week 7
Population: Number of participants analyzed = participants with EASI score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
Participants | 2 | 23

10. Secondary Outcome: Number of Patients Achieving 50% or Greater Reduction in SCORAD Score at Week 7
Description: Calculated as per description in Outcome 8.
Time Frame: Group A: Week 4; Group B: Week 7
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
Participants | 1 | 21

11. Secondary Outcome: Change in Patient Oriented Eczema Measure (POEM) Scores From Baseline to Week 7.
Description: POEM is a 7-item patient-reported quality of life outcome measure based on a questionnaire to determine disease symptoms, including bleeding, cracking, dryness, flaking, itching, sleep loss and weeping. The scoring range is from 0 to 28 (no disease to most severe disease, respectively).
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with POEM score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 17.3 [11.55 to 23.05] | 16.82 [14.26 to 19.38]
  Week 4/ Week 7 | 11.8 [6.79 to 16.81] | 5.93 [3.41 to 8.44]
  Change | 5.50 [2.90 to 8.10] | 10.89 [7.99 to 13.80]

12. Secondary Outcome: Change in Global Individual Signs Score (GISS) From Baseline to Week 7
Description: GISS assesses AD lesions for erythema, excoriations, lichenification and edema/papulation. Each component will be rated on a global basis (over the entire body surface rather than region) using a 4-point scale (0=none, 1=mild, 2=moderate and 3=severe) according to the EASI grading severity. Total score will range from 0 to 12 (no disease to most severe disease, respectively).
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with GISS score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 8.4 [6.92 to 9.88] | 9.64 [9.03 to 10.25]
  Week 4/ Week 7 | 7.5 [5.36 to 9.64] | 4.36 [3.23 to 5.48]
  Change | 0.9 [-0.19 to 1.99] | 5.28 [3.99 to 6.58]

13. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) From Baseline to Week 7
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on QOL. The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 questions, which assess QOL over the past week, with an overall scoring system of 0 to 30; a high score is indicative of a poor QOL.
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with DLQI score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 11.8 [7.18 to 16.42] | 12.93 [10.11 to 15.75]
  Week 4/ Week 7 | 6.1 [1.99 to 10.21] | 4.00 [1.43 to 6.57]
  Change | 5.70 [1.90 to 9.50] | 8.93 [6.15 to 11.70]

14. Secondary Outcome: Change in HADS (Anxiety) Score From Baseline to Week 7
Description: The HADS is a set of fourteen questions to be rated by a patient on a four point (0-3) response category so the possible scores range from 0 to 21 for anxiety and 0 to 21 for depression. Scoring is as follows:
  (0-7)= Normal (8-10)= Borderline Abnormal (11-21)= Abnormal
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: Number of participants analyzed = participants with HADS score assessment at specified time-points. Missing values imputed by LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 4.6 [2.41 to 6.79] | 7.29 [5.2 to 9.37]
  Week 4/ Week 7 | 3.2 [1.02 to 5.38] | 2.64 [1.35 to 3.93]
  Change | 1.40 [0.43 to 2.37] | 4.65 [2.84 to 6.45]

15. Secondary Outcome: Change in HADS (Depression) Score From Baseline to Week 7
Description: as for outcome 14
Time Frame: Group A: Baseline to Week 4; Group B: Baseline to Week 7
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group A: 200 mg Cohort | Group B: 400 mg Cohort
Number analyzed (Participants) | 10 | 28
score on a scale
  Baseline | 5.6 [1.59 to 9.61] | 7.11 [5.25 to 8.97]
  Week 4/ Week 7 | 4.2 [-0.98 to 9.38] | 3.18 [1.98 to 4.38]
  Change | 1.40 [-0.19 to 2.99] | 3.93 [2.35 to 5.51]

ADVERSE EVENTS:
Time Frame: Baseline to Week 7
Description: All the Adverse Events that the subjects experienced from Visit 1 Day 1 (Post-injection) until 7 days after the last administration of the study drug were captured in the clinical database. The severity of adverse events was assigned using CTCAE version 4.03.
Arm/Group | 200 mg Cohort | 400 mg Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/28
Other Adverse Events (participants affected / at risk) | 3/10 | 6/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Cohort (N=10) | 400 mg Cohort (N=28)
Site injection erythema (General disorders) | 1 (2) | 0 (0) — Grade 1 AE
site injection redness (General disorders) | 0 (0) | 2 (4) — Grade 1 AE
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1 AE
Asymptomatic sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) — Grade 1 AE
Bilateral Peripheral Edema in lower extremities (General disorders) | 0 (0) | 1 (1) — Grade 2 AE
Facial swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 1 AE
Inguinal Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1 AE
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — Grade 1 AE
Swelling on right hand (General disorders) | 0 (0) | 1 (1) — Grade 1 AE
Urinary Track Infection (Infections and infestations) | 0 (0) | 1 (1) — Grade 1 AE
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1 AE
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) — Grade 1 AE
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Grade 2 AE
worsening hypertension (Cardiac disorders) | 1 (3) | 0 (0) — Grade 2 AE
worsening hypertension (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3 AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution shall provide the Sponsor a copy of each proposed publication, abstract or presentation at least ninety days in advance for a proposed publication to a journal, editor or other third party. The Sponsor shall, within sixty days, advise Institution if there is any of the Sponsor's Confidential Information in proposed publication. Institution shall delete any of the Sponsor's Confidential Information prior to submitting and/or presenting.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03496974/Prot_SAP_000.pdf